CLINICAL TRIAL: NCT00335400
Title: Comparison of an Anesthetic and Dilating Gel Cocktail Versus the Standard Pre-operative Pharmacologic Regimen for Cataract Surgery on Corneal Anesthesia and Pupil Dilation.
Brief Title: Anesthetic and Dilating Gel for Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Sherif R El-Defrawy, Principal Investigator, Queen's University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QUEENS-SRE-1
Record Dates: First submitted 2006-06-08; First posted 2006-06-09 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

INTERVENTIONS:
Drug: Anesthetic Dilating Gel

SUMMARY:
To prepare the eye for cataract surgery, drugs must be given to the eye to allow for surgery to take place. Traditionally, dilating drops and drops containing NSAIDs (to control inflammation) are given to the patient well in advance of surgery at repeated time intervals. As well, a gel containing lidocaine is applied to the eye just prior to surgery to anesthetize (reduce pain and feeling) in the area of the eye. Although effective, the procedure is time-consuming and costly for nursing staff. Recently, a few hospitals have reported success in mixing the pupil-dilating and NSAID drops with the lidocaine gel, creating an "anesthetic dilating gel". Although success has been reported, there have been no studies to clearly demonstrate that the "anesthetic dilating gel" is as effective at dilating the pupil and reducing sensitivity of the cornea during surgery than the traditional methods of drops and gel. It is possible that the dilating gel is less effective due to slower diffusion of drugs into the eye. The study will compare the effectiveness of the anesthetic dilating gel with the standard pre-operative pharmacologic regimen for cataract surgery. Stability (maintaining effectiveness over time) and contamination of the study gel will also be assessed. If the dilating gel is shown to be as effective in regards to pupil dilation and corneal anesthesia, while maintaining stability and sterility over time, hospitals can be encouraged to use such a anesthetic dilating gel routinely during pre-operative procedures before cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for first cataract surgery (i.e., first eye)

Exclusion Criteria:

* previous ocular surgery,
* pseudoexfoliation syndrome,
* diabetes,
* herpetic eye disease,
* posterior synechiae,
* previous uveitis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-03; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Pupil dilation
Corneal anesthesia

SECONDARY OUTCOMES:
Gel stability
Gel sterility
Patient comfort

CONTACTS AND LOCATIONS:
Overall Officials: Sherif El-Defrawy, MD PhD FRCSC, Principal Investigator — Hotel Dieu Hospital, Kingston General Hospital, Queen's University
Locations (1):
- Hotel Dieu Hospital, Kingston, Ontario, Canada